CLINICAL TRIAL: NCT05222542
Title: Angiotensin Metabolite Profile After Subarachnoid Hemorrhage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Roman Ullrich (Other)
Collaborators: Austrian Science Fund (FWF) (Other)
Responsible Party: Sponsor-Investigator, Dr. Roman Ullrich, Prof., sub-investigator, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: EK Nr: 1681/2021
Record Dates: First submitted 2022-01-11; First posted 2022-02-03 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
Keywords: Cerebral vasospasm; Renin angiotensin system
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma (without DNA) and cerebrospinal fluid (potentially containing cellular residues with DNA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients after aneurysmal subarachnoid hemorrhage: Samples (plasma, and in patients with in-dwelling cerebrospinal fluid drainages also cerebrospinal fluid) will be taken within 72 hours of subarachnoid hemorrhage and 7, 14 and 21 days following initial bleeding. Another plasma sample will be obtained if an antihypertensive therapy with a RAS modifying drug has been started.
  Interventions: Other: Sampling of plasma and cerebrospinal fluid at specified time points

INTERVENTIONS:
Other: Sampling of plasma and cerebrospinal fluid at specified time points — Samples (plasma, and in patients with in-dwelling cerebrospinal fluid drainages also cerebrospinal fluid) will be taken within 72 hours of subarachnoid hemorrhage and 7, 14 and 21 days following initial bleeding. Another plasma sample will be obtained if an antihypertensive therapy with a RAS modifying drug has been started.

SUMMARY:
The outcome of subarchnoid hemorrhage depends on the severity of the bleeding and the development of secondary neurologic deficits caused by cerebral vasospasm. The primary endpoint is a comparison of renin angiotensin system (RAS) parameters (plasma concentrations of Angiotensin [Ang] I, Ang II, Ang 1-7, and Ang 1-5, angiotensin metabolite based markers of RAS enzyme activities as well as active ACE and ACE2 concentrations in plasma and CSF) between patients with and without vasospasm, mechanical ventilation, antihypertensive therapy with a RAS modifying drug and low versus high Hunt and Hess grade of subarachnoid hemorrhage.

DETAILED DESCRIPTION:
Wider research context. The clinical course and neurological outcome of patients with subarachnoid hemorrhage following rupture of an intracranial aneurysm depend on surgical repair of the ruptured aneurysm to avoid rebleeding and the development of cerebral vasospasm that may cause delayed ischemic deficits. Up to 65% of patients require mechanical ventilation mostly due to neurologic deficits or hypoxia. The renin angiotensin system (RAS) is acutely activated after subarachnoid hemorrhage with increased renin and angiotensin (Ang) II plasma levels, but effects of the vasoconstrictor Ang II on development of vasospasm have not been investigated in patients. The RAS may also be activated by mechanical ventilation, but it is unknown if this has an impact on occurrence of vasospasm. Arterial hypertension is an important risk factor for subarachnoid hemorrhage and vasospasm, and around 50% of patients have a history of high blood pressure. During weaning from mechanical ventilation arterial hypertension is a wide spread clinical problem, but how RAS modifying drugs act on the angiotensin metabolite profile that may already be dysregulated after subarachnoid hemorrhage remains unclear.

Objectives. To investigate associations between angiotensin metabolite profile (Ang I, Ang II, Ang 1-7 and Ang 1-5 concentrations) and angiotensin converting enzyme (ACE) and ACE2 activities in plasma as well as ACE and ACE2 activities in cerebrospinal fluid (CSF) and development of cerebral vasospasm in patients with and without mechanical ventilation following subarachnoid hemorrhage, and to find out how the angiotensin metabolite profile is changed by antihypertensive therapy with a RAS modifying drug in these patients.

Methods. Ang I, Ang II, Ang 1-7 and Ang 1-5 equilibrium concentrations will be measured by liquid chromatography tandem mass spectrometry in 60 patients after subarachnoid hemorrhage in plasma. Active ACE and ACE2 concentrations will be measured in plasma and in CSF in patients with CSF drainages. Samples will be taken within 72 hours of subarachnoid hemorrhage and 7, 14 and 21 days following initial bleeding. Another plasma sample will be obtained if an antihypertensive therapy with a RAS modifying drug has been started. Angiotensin metabolite based markers of RAS enzyme activities will be calculated for renin and ACE activities and alternative RAS activation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of subarachnoid hemorrhage because of aneurysmal rupture admitted to the ICU
* Invasive monitoring of arterial blood pressure

Exclusion Criteria:

* Patients who decline study participation
* Brain stem death
* Chronic renal impairment with creatinine > 2mg/dL or hemodialysis
* Chronic liver failure of Child Pugh class C or higher
* Chronic heart failure
* Hormone producing neuroendocrine tumor
* Sarcoidosis
* Pregnancy
* Planned transfer to another hospital shortly after aneurysm repair

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of subarachnoid hemorrhage because of aneurysmal rupture admitted to the ICU
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Angiotensin metabolite concentrations within 72 hours | within 72 hours of subarachnoid hemorrhage
  Ang I, Ang II, Ang 1-7 and Ang 1-5 equilibrium concentrations in plasma (in pmol/L), comparison between patients with and without vasospasm, with and without mechanical ventilation and low versus high Hunt and Hess grade
Angiotensin metabolite concentrations after 7 days | 7 days after subarchnoid hemorrhage
  Ang I, Ang II, Ang 1-7 and Ang 1-5 equilibrium concentrations in plasma (in pmol/L), comparison between patients with and without vasospasm, with and without mechanical ventilation and low versus high Hunt and Hess grade
Angiotensin metabolite concentrations after 14 days | 14 days after subarchnoid hemorrhage
  Ang I, Ang II, Ang 1-7 and Ang 1-5 equilibrium concentrations in plasma (in pmol/L), comparison between patients with and without vasospasm, with and without mechanical ventilation and low versus high Hunt and Hess grade
Angiotensin metabolite concentrations after 21 days | 21 days after subarchnoid hemorrhage
  Ang I, Ang II, Ang 1-7 and Ang 1-5 equilibrium concentrations in plasma (in pmol/L), comparison between patients with and without vasospasm, with and without mechanical ventilation and low versus high Hunt and Hess grade
ACE concentrations within 72 hours | within 72 hours of subarachnoid hemorrhage
  active ACE concentrations in plasma and cerebrospinal fluid (in µg/mL), comparison between patients with and without vasospasm, with and without mechanical ventilation and low versus high Hunt and Hess grade
ACE concentrations after 7 days | 7 days after subarachnoid hemorrhage
  active ACE concentrations in plasma and cerebrospinal fluid (in µg/mL), comparison between patients with and without vasospasm, with and without mechanical ventilation and low versus high Hunt and Hess grade
ACE concentrations after 14 days | 14 days after subarachnoid hemorrhage
  active ACE concentrations in plasma and cerebrospinal fluid (in µg/mL), comparison between patients with and without vasospasm, with and without mechanical ventilation and low versus high Hunt and Hess grade
ACE concentrations after 21 days | 21 days after subarachnoid hemorrhage
  active ACE concentrations in plasma and cerebrospinal fluid (in µg/mL), comparison between patients with and without vasospasm, with and without mechanical ventilation and low versus high Hunt and Hess grade
ACE2 concentrations within 72 hours | within 72 hours of subarachnoid hemorrhage
  active ACE2 concentrations in plasma and cerebrospinal fluid (in ng/mL), comparison between patients with and without vasospasm, with and without mechanical ventilation and low versus high Hunt and Hess grade
ACE2 concentrations after 7 days | 7 days after subarachnoid hemorrhage
  active ACE2 concentrations in plasma and cerebrospinal fluid (in ng/mL), comparison between patients with and without vasospasm, with and without mechanical ventilation and low versus high Hunt and Hess grade
ACE2 concentrations after 14 days | 14 days after subarachnoid hemorrhage
  active ACE2 concentrations in plasma and cerebrospinal fluid (in ng/mL), comparison between patients with and without vasospasm,with and without mechanical ventilation and low versus high Hunt and Hess grade
ACE2 concentrations after 21 days | 21 days after subarachnoid hemorrhage
  active ACE2 concentrations in plasma and cerebrospinal fluid (in ng/mL), comparison between patients with and without vasospasm, with and without mechanical ventilation and low versus high Hunt and Hess grade
Impact of RAS modifying drugs after subarachnoid hemorrhage | after start of a RAS modifying drug therapy for arterial hypertension in the intensive care unit
  Ang I, Ang II, Ang 1-7 and Ang 1-5 equilibrium concentrations in plasma (in pmol/L), comparison between sample taken after start of a RAS modifying drug and the previous sample in the study schedule

SECONDARY OUTCOMES:
Correlation of RAS analyses with clinical parameters | Within 72 hours, 7, 14 and 21 days following subarachnoid hemorrhage and after start of a RAS modifying drug therapy for arterial hypertension in the intensive care unit
  Correlations of RAS parameters (Ang I, Ang II, Ang 1-7 and Ang 1-5 equilibrium concentrations and active ACE and ACE2 concentrations) and aldosterone plasma concentrations with blood pressure, blood pressure target, routine laboratory parameters and ventilator settings, and comparison of RAS parameters and aldosterone plasma concentrations between men and women

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Krenn, MD, PhD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
The data will be shared and made accessible after publishing of the results of the study according to the European code of conduct for research integrity - as open as possible and as closed as necessary. Results will be published in an accurate, transparent manner in an international peer reviewed journal supporting open access. As persistent identifier DOI will be used.